CLINICAL TRIAL: NCT07278830
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Safety and Efficacy of Recombinant Fully Human Anti-PCSK9 Monoclonal Antibody Injection (SAL003) Combined With Atorvastatin in Subjects With Hypercholesterolemia and Mixed Dyslipidemia
Brief Title: A Phase II Study to Evaluate the Safety and Efficacy of SAL003 Combined With Atorvastatin in Hypercholesterolemia and Mixed Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Salubris (Chengdu) Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL003A201
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Hypercholesterolemia and Mixed Dyslipidemia
Keywords: LDL-C (Low-Density Lipoprotein Cholesterol); PCSK9 Inhibitor; SAL003
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group Q4W (Experimental)
  Interventions: Drug: SAL003 140mg+Atorvastatin
- Test Group Q8W (Experimental)
  Interventions: Drug: SAL003 420mg+Atorvastatin
- Reference Group Q4W (Placebo Comparator)
  Interventions: Drug: Placebo 140mg+Atorvastatin
- Reference Group Q8W (Placebo Comparator)
  Interventions: Drug: Placebo 420mg+Atorvastatin

INTERVENTIONS:
Drug: SAL003 140mg+Atorvastatin — Double-blind treatment period: During the stable dose of atorvastatin treatment, 140mg of SAL003 was administered once every 4 weeks for a total of 6 times. Extended treatment period: During the stable dose of atorvastatin treatment, 140mg of SAL003 was administered once every 4 weeks for a total of 2 times.
  Arms: Test Group Q4W
Drug: SAL003 420mg+Atorvastatin — Double-blind treatment period: During the stable dose of atorvastatin treatment, 420mg of SAL003 was administered once every 8 weeks for a total of 3 times. Extended treatment period: During the stable dose of atorvastatin treatment, 140mg of SAL003 was administered once every 4 weeks for a total of 2 times.
  Arms: Test Group Q8W
Drug: Placebo 140mg+Atorvastatin — Double-blind treatment period: During the stable dose of atorvastatin treatment, 140mg of Placebo was administered once every 4 weeks for a total of 6 times. Extended treatment period: During the stable dose of atorvastatin treatment, 140mg of SAL003 was administered once every 4 weeks for a total of 2 times.
  Arms: Reference Group Q4W
Drug: Placebo 420mg+Atorvastatin — Double-blind treatment period: During the stable dose of atorvastatin treatment, 420mg of Placebo was administered once every 8 weeks for a total of 3 times. Extended treatment period: During the stable dose of atorvastatin treatment, 140mg of SAL003 was administered once every 4 weeks for a total of 2 times.
  Arms: Reference Group Q8W

SUMMARY:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of SAL003, a recombinant fully human anti-PCSK9 monoclonal antibody, in combination with a stable dose of atorvastatin in patients with hypercholesterolemia and mixed dyslipidemia.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy, safety, and pharmacokinetics of SAL003, a recombinant fully human anti-PCSK9 monoclonal antibody, when used in combination with stable, background atorvastatin therapy in adult patients with hypercholesterolemia and mixed dyslipidemia.

The study is structured into four distinct periods to ensure patient eligibility, standardize background therapy, and assess both short-term and longer-term effects of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 to 75 years.
2. Diagnosis of hypercholesterolemia and/or mixed dyslipidemia per the 2016 Chinese guidelines.
3. On a stable statin regimen as defined by the two pathways:

   * Pathway 1: On other statins or irregular atorvastatin, willing to switch to/stabilize on atorvastatin.
   * Pathway 2: On stable, regular atorvastatin (Lipitor) for ≥4 weeks.
4. Fasting LDL-C must be above target:

   * With ASCVD history: ≥1.8 mmol/L (70 mg/dL)
   * Without ASCVD history: ≥2.6 mmol/L (100 mg/dL)
5. Fasting triglycerides (TG) ≤ 5.6 mmol/L (500 mg/dL) at screening.
6. Provide signed informed consent.

Exclusion Criteria:

1. Suffering from homozygous familial hypercholesterolemia (HoFH); Other diseases that may cause secondary increase of LDL-C: Cushing's syndrome, nephrotic syndrome, myeloma, glycogen storage disease, systemic lupus erythematosus, acute intermittent porphyria;
2. Route 1: The medication compliance of atorvastatin during the induction period is less than 80% or more than 120%; Route 2: The medication compliance of atorvastatin within 28 days before screening is less than 80% or more than 120%;
3. Within 3 months before screening, there is heart failure (NYHA cardiac function classification of grade III and IV), acute coronary syndrome, percutaneous coronary intervention, or other serious heart diseases [such as cardiogenic shock, grade II-III atrioventricular block, bradycardia (heart rate < 50 beats/minute), other serious arrhythmias, etc.];
4. Within 3 months before screening, there is a serious cerebrovascular disease (hypertensive encephalopathy, cerebral vascular injury, stroke, transient ischemic attack, etc.), or there is a serious aortic or peripheral vascular lesion, or there are indications for surgical intervention;
5. Within 3 months before screening, there is a major surgical history or plans to undergo major surgery during the study period;
6. Patients with poorly controlled hypertension (SBP ≥ 160 mm Hg or DBP ≥ 100 mm Hg);
7. Diabetic patients with the following conditions known: 1) Type 1 diabetic patients; 2) Type 2 diabetic patients with poor blood sugar control (HbA1c > 8.0%);
8. Patients with active viral hepatitis (including hepatitis B and hepatitis C), other severe liver diseases, or liver dysfunction (ALT or AST > 2.5 times the upper limit of normal, TBIL > 2 times the upper limit of normal);
9. Glomerular filtration rate (eGFR) < 30 ml/min/1.73m2 during the screening period;
10. Patients with abnormal thyroid function (thyroid stimulating hormone TSH exceeds the normal range of the center);
11. CK > 3 times the upper limit of normal during the screening period;
12. Positive for AIDS or syphilis tests;
13. Active malignant tumors, or patients with a history of malignant tumors within 5 years before screening (excluding skin basal cell carcinoma or cervical carcinoma in situ);
14. Patients known to be allergic to the test drug or any component of the test drug, or who have had a severe allergic reaction to other antibody-based drugs;
15. Patients with a history of organ transplantation;
16. Within 3 months before screening, blood donation or significant blood loss (> 400 mL), or those diagnosed with insufficient blood volume;
17. Within 30 days before the administration of the study drug, use of any known substances that can affect lipid metabolism, tonics (such as fish oil > 1000 mg/day, drugs containing red yeast rice components or health supplements), or other cholesterol-lowering drugs other than statins;
18. Within 3 months before screening, participated in other drug or device clinical trials, or within 6 months before screening received any treatment targeting the proprotein convertase subtilisin/kexin type 9 (PCSK9) target;
19. Within 6 months before screening had a history of drug abuse or alcoholism (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
20. Female subjects during the screening period or during the trial are breastfeeding or have a positive serum pregnancy result;
21. The subject or the subject's spouse or partner has a pregnancy plan or refuses to adopt an acceptable effective contraceptive method from the time of signing the informed consent form to the end of the last administration;
22. The subject and his/her spouse or partner have a pregnancy plan or refuse to adopt an acceptable effective contraceptive method from the time of signing the informed consent form to the end of the last administration within 6 months;
23. Patients considered not suitable for participating in the clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Percent change of Low-Density Lipoprotein Cholesterol (LDL-C) | at Week 24
  Percent change from baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University，Guangzhou，Guangdong，510120, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No